CLINICAL TRIAL: NCT03357029
Title: Neuromodulation in Patients With Painful Chronic Pancreatitis - A Randomized, Double-blind, Sham-controlled, Prospective, Cross-over, Controlled Study in Chronic Pain Investigating if a Novel Vagal Neuromodulation Approach Provides Analgesic Benefit Through Central Mechanisms in Patients With Chronic Pancreatitis
Brief Title: Neuromodulation in Patients With Painful Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Brøndum Frøkjær (Other)
Collaborators: ElectroCore INC (Industry)
Responsible Party: Sponsor-Investigator, Jens Brøndum Frøkjær, MD, Professor, PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VNS project
Record Dates: First submitted 2017-11-21; First posted 2017-11-29 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Painful Chronic Pancreatitis; Visceral Pain; Neuropathic Pain
Keywords: Chronic pancreatitis; Vagal nerve stimulation; Visceral Pain
MeSH Terms: conditions — Visceral Pain; Neuralgia; Pancreatitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Gammacore Device (Active Comparator): The GammaCore Device is a non-Invasive vagus nerve stimulator. One stimulation dose bilaterally to the cervical vagal neck area, three times per day (morning 8 am., afternoon 2 pm, and evening 8 pm) for two weeks
  Interventions: Device: GammaCore Device
- Sham Device (Sham Comparator): The Sham GammaCore device looks and operates like the Active GammaCore device, but does not deliver a therapeutic stimulation treatment.
  One stimulation dose bilaterally to the cervical vagal neck area, three times per day (morning 8 am., afternoon 2 pm, and evening 8 pm) for two weeks.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: GammaCore Device — GammaCore will be administered using a handheld device the size of a mobile phone, which consists of a battery powered portable stimulator with a digital control user interface that controls the stimulation amplitude and two steel contact electrodes.
  Arms: Gammacore Device
Device: Sham Device — Sham device will be administered using a handheld device the size of a mobile phone, which consists of a battery powered portable stimulator with a digital control user interface that controls the stimulation amplitude and two steel contact electrodes. The sham device is identical in appearance, weight, visual and audible feedback, and user application and control but did not deliver electrical stimulations.
  Arms: Sham Device

SUMMARY:
The purpose of this trial is to explore if a novel vagal neuromodulation approach provides analgesic benefit through central mechanisms in patients with chronic pancreatitis

DETAILED DESCRIPTION:
This study is a randomized, double blind, sham-controlled, cross-over, controlled investigation. The overall objective of the study is to conduct a study of vagal tone and the sensory system (brain activity, sensory testing, and questionnaires) assessing the effect of two weeks' transcutaneous vagal neuromodulation in chronic pancreatitis patients not responding adequately to traditional pharmacological pain treatment, in comparison to the effect of two weeks' sham treatment. The active treatment will be performed using a commercially available and validated device called GammaCore (the active treatment) while the sham treatment will be performed using a sham-device. GammaCore device is a non-invasive neurostimulator that has been approved for the treatment of anxiety, primary headache, including migraine.

The study will begin with a one-week baseline registration period, in which the patients will receive no treatment. Next, the baseline period will be followed by a 2-week treatment period where the subjects will be randomized to either active treatment or the sham treatment. Afterwards, a wash-out period of one week and a second baseline registration period of one week will occur. Finally, in the second treatment period the patients will switch in treatment assignment, meaning that patient who received active treatment in the beginning, will now receive sham treatment and vice versa. During both treatments, the patients will be asked to self-administer one stimulation dose bilaterally to the cervical vagal neck area, three times per day (morning 8 am., afternoon 2 pm, and evening 8 pm). During the whole study, subjects will be asked to complete a pain diary and several questionnaires. Moreover, at the beginning and end of each treatment period (four times), all subjects will undergo testing which will include magnetic resonance imaging (MRI), quantitative sensory testing (QST), cardiac vagal tone (CVT) and collecting blood samples.

The primary efficacy parameters to be evaluated are clinical pain relief and brain alterations using MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the ages of 18 with a diagnosis of CP diagnosed using the Mayo Clinic diagnostic criteria.
* The participants must be able to read and understand Danish.
* The patients must suffer from chronic abdominal pain characteristic for CP, meet the criteria for chronic pain (pain ≥ 3 days per week in at least 3 months) and must consider their pain as insufficiently treated with their usual analgesic treatment.
* Personally, signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial as well as signing the following document: "Informeret samtykke om opbevaring af biologisk material i biobank til fremtidig forskning".
* Personally, signed and dated the Power of attorney document (Fuldmagtserklæring) indicating that the patient has accepted that the Danish Medical Agency Sundhedsstyrelsen/Lægemiddelstyrelen) have access to the medical records.
* Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other trial procedures.

Exclusion Criteria:

* Patients with any clinically significant abnormalities that in the opinion of the investigator may increase the risk associated with trial participation or may interfere with the interpretation of the trial results.
* Alcohol dependence (Alcohol use in accordance with the recommendations by the Danish Health and Medicines Authority are allowed).
* Illegal drug dependencies.
* Participating in another study where investigational drug is used.
* Patients must not suffer from painful conditions other than CP that make them unable to distinguish the pain associated with CP from chronic pain of other origin.
* Cardiovascular diseases
* Low blood pressure < 100/60
* Not able to understand or follow the instructions.
* Any condition with elevated intracranial pressure.
* Female patients who are pregnant or lactating, or intend to become pregnant and male patients who intend to father a child during the course of the study. A pregnancy test will be conducted at baseline and after 8 weeks to ensure that female patients are not pregnant during the study medication period. The investigator will have to urge that fertile female patients use a safe contraception method during the study and for at least 15 hours after termination of the study medication period. The following methods are considered as safe contraception methods:

  * The combined oral contraceptive pill
  * Intra uterine device
  * Gestagen injection
  * Subdermal implantation
  * Hormone vaginal ring
  * Transdermal plaster
* Contraindications for MRI: Such as metallic Foreign Body in the Eye, "Triggerfish" Contact Lens, Gastric Reflux Device, Insulin Pumps, Permanent pacemaker, Temporary external transvenous pacing leads, Other implantable metallic components which is considered unsafe by the medical doctor.
* Previous surgery on vagus nerve.
* Known neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The perceived clinical pain measured by pain diary based on Visual Analog Scale (VAS) | Up to 8 weeks.
  The primary clinical efficacy parameter to be evaluated is pain relief. In the clinical part of the study the efficacy is assessed as changes in the daily experience of pain, which will be measured using a patient pain diary based on the visual analog scale (VAS). Maximum intensity and average daily VAS will be recorded on daily basis.
Detection of brain changes using magnetic resonance imaging (MRI) | Up to 8 weeks.
  The primary experimental endpoint is detection of structural, functional, metabolic brain alterations using MRI techniques in order to study the brain mechanisms involved in chronic pain and central sensitization.

SECONDARY OUTCOMES:
Change in quality of life QoLQ | Up to 8 weeks.
Changes in pain and physical functioning composite scores of the modified brief pain inventory-short form (mBPI-sf). | Up to 8 weeks.
Patient Global Impression of Change (PGIC). | Up to 8 weeks.
Quantitative sensory testing (thermal, mechanical and muscle stimulation, including conditioned pain modulation) | Up to 8 weeks.
Cardiac vagal tone | Up to 8 weeks.
Blood samples | Up to 8 weeks.
  Changes in cytokines will be assessed .

CONTACTS AND LOCATIONS:
Locations (1):
- Mech-Sense, Department of Radiology, Aalborg, Denmark

REFERENCES:
- [Derived] Muthulingam JA, Olesen SS, Hansen TM, Brock C, Drewes AM, Frokjaer JB. Cervical transcutaneous vagal neuromodulation in chronic pancreatitis patients with chronic pain: A randomised sham controlled clinical trial. PLoS One. 2021 Feb 26;16(2):e0247653. doi: 10.1371/journal.pone.0247653. eCollection 2021. PMID 33635894
- [Derived] Muthulingam JA, Olesen SS, Hansen TM, Brock C, Drewes AM, Frokjaer JB. Study protocol for a randomised double-blinded, sham-controlled, prospective, cross-over clinical trial of vagal neuromodulation for pain treatment in patients with chronic pancreatitis. BMJ Open. 2019 Aug 23;9(7):e029546. doi: 10.1136/bmjopen-2019-029546. PMID 31603076